CLINICAL TRIAL: NCT03775356
Title: Reduction of Intraoperative EEG Burst Suppression - Test of Efficacy
Brief Title: Reduction of Intraoperative EEG Burst Suppression
Acronym: BsR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BsR
Record Dates: First submitted 2018-11-22; First posted 2018-12-13 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2020-09

CONDITIONS: Burst Suppression; EEG With Abnormally Slow Frequencies; Postoperative Delirium
Keywords: Intraoperative EEG based monitoring; Level of hypnosis; Burst suppression; Postoperative delirium; EEG-signal characteristics; Entropy
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Single masked. The entropy and EEG module will be masked for the responsible anesthetist as well as the study team during the entire investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - Blinded (No Intervention): EEG and Entropy will be blinded. The anesthesiological management will be performed by the anesthetist according to clinical standard operations.
- 2 - Unblinded (Active Comparator): EEG and Entropy will be unblinded. The intervention starts with the start of a positive burst suppression rate. In the case of a concurrent hypotension the anesthetist treats the hypotension according to clinical standard operations in the first step. Hypotension means blood pressure values blow the baseline value which is defined by the lowest, preoperatively measured value. If after this treatment and a reevaluation of the BSR, BSR remains positive, the anesthetist is going to reduce the concentration of anesthetics in a second step. In case of positive BSR and a blood pressure value ≥ the baseline value, the concentration of anesthetics will be reduced as a first measure. The aim is to figure out whether one or both of these interventions can reduce to total, cumulative BSR.
  Interventions: Other: Treatment of hypotension and/or reduction of anesthetics

INTERVENTIONS:
Other: Treatment of hypotension and/or reduction of anesthetics — The treatment of hypotension can be done by the responsible anesthetist according to the clinical standard operations including any accepted drug typically used in this hospital. The reduction of anesthetics can be done either by reducing the volatile end tidal anesthetics concentration (ETAC) or the infusion rate of propofol.
  Arms: 2 - Unblinded

SUMMARY:
Burst suppression (BS) is a not physiological pattern in the electroencephalogram (EEG). BS during general anesthesia is mainly seen as a sign for too deep hypnosis and may increase the risk of postoperative delirium (POD), a disturbance of consciousness arising within 24 hours after surgery. This monocentric, simple masked randomized study aims primarily to investigate, whether particular anesthesiological interventions reduce the occurrence of intraoperative burst suppression. The investigator initiated trial includes 66 patients (male and female) aged ≥ 60 years in two groups (intervention and control group). Secondary aims will be the correlation of burst suppression and mean arterial pressure, concentration of anesthetics and postoperative delirium.

DETAILED DESCRIPTION:
Intraoperative burst suppression represents a non physiological EEG pattern. According to the literature and scientific knowledge, intraoperative burst suppression patterns might be caused either by hypotension resulting in a reduced cerebral circulation or by an oversedation of anesthetics correlating with a very deep level of hypnosis.

Some publications exist that discuss the occurrence of intraoperative burst suppression especially in elderly people (aged ≥ 60 years) as a predictor of postoperative delirium and postoperative cognitive dysfunction.

None of the studies however was able to prove a causal relationship between burst suppression and postoperative delirium. Contrary it might simply be an epiphenomenon.

Conducting this interventional trail primarily aims to prove whether specific anesthesiological interventions, such as the treatment of intraoperative hypotension in first line and/or the reduction of the concentration of anesthetics in second line, reduce intraoperative burst suppression. Hence it might be possible to investigate a possible casualty between burst suppression and postoperative delirium in a second trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Surgical interventions in general anesthesia (volatile or total intravenous anesthesia)
* expected surgery duration ≥ 1h
* American Society of Anesthesiologists (ASA) 1-4
* written informed consent prior to study participation

Exclusion Criteria:

* Neurological or psychiatric disorders
* hearing difficulty
* deafness
* neurosurgical (intra)cranial surgery
* pregnancy
* expected continuous mandatory ventilation after surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Chance of the total, cumulative burst suppression rate. | During general anesthesia and within the intervention
  The total, cumulative burst suppression rate (BSR) corresponds to area under the curve and is defined by the BSR (%) and the absolute duration of BSR (t).

SECONDARY OUTCOMES:
Burst suppression rate during induction. | During induction within the intervention
  Rate of change of the burst suppression rate during induction.
Burst suppression rate during maintenance. | During maintenance within the intervention
  Rate of change of the burst suppression ratio during maintenance.
Mean arterial blood pressure. | During burst suppression within general anesthesia
  Evaluation of the mean arterial blood pressure with positive burst suppression rate.
Endtidal anesthetic concentration (ETAC) and infusion rate of propofol. | During burst suppression within the intervention
  Evaluation of the mean ETAC and infusion rate of propofol.
Specific characteristics of the EEG frequency spectrum during burst suppression | During burst suppression within general anesthesia
  Evaluation of specific EEG frequencies differentiating BSR caused by hypotension or oversedation of anesthetics.
Postoperative delirium. | Within the first three postoperative days
  Screening of the patients regarding a postoperative delirium by a brief confession assessment method (bCAM).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schneider, Prof. Dr., Principal Investigator — Clinic director - Department of anesthesiology and intensive care
Locations (1):
- Klinikum rechts der Isar - Klinik fuer Anaesthesiologie und Intensivmedizin, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Sessler DI, Sigl JC, Kelley SD, Chamoun NG, Manberg PJ, Saager L, Kurz A, Greenwald S. Hospital stay and mortality are increased in patients having a "triple low" of low blood pressure, low bispectral index, and low minimum alveolar concentration of volatile anesthesia. Anesthesiology. 2012 Jun;116(6):1195-203. doi: 10.1097/ALN.0b013e31825683dc. PMID 22546967
- [Derived] Schussler J, Ostertag J, Georgii MT, Fleischmann A, Schneider G, Pilge S, Kreuzer M. Preoperative characterization of baseline EEG recordings for risk stratification of post-anesthesia care unit delirium. J Clin Anesth. 2023 Jun;86:111058. doi: 10.1016/j.jclinane.2023.111058. Epub 2023 Jan 25. PMID 36706658
- [Derived] Fleischmann A, Georgii MT, Schuessler J, Schneider G, Pilge S, Kreuzer M. Always Assess the Raw Electroencephalogram: Why Automated Burst Suppression Detection May Not Detect All Episodes. Anesth Analg. 2023 Feb 1;136(2):346-354. doi: 10.1213/ANE.0000000000006098. Epub 2022 Jun 2. PMID 35653440
- [Derived] Georgii MT, Kreuzer M, Fleischmann A, Schuessler J, Schneider G, Pilge S. Targeted Interventions to Increase Blood Pressure and Decrease Anaesthetic Concentrations Reduce Intraoperative Burst Suppression: A Randomised, Interventional Clinical Trial. Front Syst Neurosci. 2022 Mar 4;16:786816. doi: 10.3389/fnsys.2022.786816. eCollection 2022. PMID 35308563